CLINICAL TRIAL: NCT04546503
Title: Evaluation of the Interest of Regional Locoregional Anesthesia by Perfusion Blocks in Continuous Infusion in Polytrauma Patients With Limb Fractures and Mechanical Ventilation. A Prospective Randomized Study
Brief Title: Impact of Continuous Regional Analgesia in Severe Trauma Patients
Acronym: ALRréa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 8822; 2010-A00443-36 (Other: ID RCB)
Record Dates: First submitted 2017-10-19; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2017-10

CONDITIONS: Limb Fracture
Keywords: Intensive Care Unit ; limb fracture ; regional analgesia
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Aseptic placement of one or two tunnelized CPNB at the level of the nerves or plexus of the traumatized limb (s), Nervestimulation and ultrasound guidance by trained operator.
  Continuous infusion of ropivacaine 0.2% at 1mL/10 Kg /H
  group with locoregional anesthesia: Sedation using midazolam and sufentanil: Multi-Daily adjustment of doses every 4 hours using Behavioral Pain Scale score <4 and Ramsay Score > 4 + peronerval block catheter from 0 to 24h after admission in intensive care unit using ropivacaine 0.2% with a continuous infusion at 1mL/10 Kg /H
Who Masked: Investigator
Masking Description: The investigator responsible for assessing sedation and adjusting dosages hypnotic and morphinic (according to objectives) will not be aware of the result of the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Regional Analgesia group (Active Comparator): Sedation using midazolam and sufentanil: Multi-Daily adjustment of doses every 4 hours using Behavioral Pain Scale score <4 and Ramsay Score > 4 + perinerval block catheter from 0 to 24h after admission in intensive care unit using ropivacaine 0.2% with a continuous infusion at 1mL/10 Kg /H
  Interventions: Procedure: Control Group
- Control Group (Experimental): group with general anesthesia and without locoregional anesthesia: Sedation using midazolam and sufentanil: Multi-Daily adjustment of doses every 4 hours using Behavioral Pain Scale score <4 and Ramsay Score > 4
  Interventions: Procedure: Continuous Regional analgesia

INTERVENTIONS:
Procedure: Continuous Regional analgesia — Aseptic placement of one or two tunnelized CPNB at the level of the nerves or plexus of the traumatized limb (s), Nervestimulation and ultrasound guidance by trained operator.
  Continuous infusion of ropivacaine 0.2% at 1mL/10 Kg /H
  + General anaesthesia
  Arms: Control Group
Procedure: Control Group — General anaesthesia without regional analgesia
  Arms: Continuous Regional Analgesia group

SUMMARY:
Regional analgesia, based on its physiological effects and efficacy, is used for optimal perioperative pain relief. However, for acute pain in multiple trauma patients in a critical condition, it has not been prospectively studied. The use of regional anaesthesia in this group of patients extend to the management of trauma patients and of other painful procedures performed at the patient's bed. The use of RA in such patients must be analyzed in the light of associated conditions that can increase the risk of systemic toxicity and complications: coagulopathies, infection, immunosuppressive states, sedation and problems associated with mechanical ventilation. The investigators aim to assess the role of continuous peripheral nerve blocks (CPNB) in multiple trauma patients, in order to show the benefits in terms of opiates consumption decrease, sedation limitation, improvement in ventilator free days and patients outcome

DETAILED DESCRIPTION:
Inclusion of multiple trauma patients with limb fractures and need for sedation and prolonged mechanical ventilation.

Patients should meet the following criterias: pressure of cerebral perfusion>60mmHg, normothermia, PaCO2 35-40 mmHg, pH> 7.20, Normal coagulation parameters, Hb> 8g / dl (without head trauma) or Hb> 10g / dl (if associated head trauma).

Randomization in two patients groups: "RA group" versus "NoRA Group

Methods:

group without locoregional anesthesia: Sedation using midazolam and sufentanil: Multi-Daily adjustment of doses every 4 hours using Behavioral Pain Scale score <4 and Ramsay Score > 4.

group with locoregional anesthesia: Sedation using midazolam and sufentanil: Multi-Daily adjustment of doses every 4 hours using Behavioral Pain Scale score <4 and Ramsay Score > 4 + peronerval block catheter from 0 to 24h after admission in intensive care unit using ropivacaine 0.2% with a continuous infusion at 1mL/10 Kg /H Follow-up up to 5 days for the 2 group. The main objective: sufentanil consumption (reported in µg / kg / d) for the same levels of Behavioral Pain Scale and Ramsay Scales values.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years
* Multiple trauma Patient ( with or without head trauma)
* Patient admitted to ICU
* Patient with limb fracture (s)
* Patient requiring sedation and mechanical ventilation for more than 48h
* Patient affiliated to a social security system
* Patient whose informed consent was obtained from the family

Exclusion Criteria:

* Patient currently enrolled in another trial
* Patient with coagulation disorders
* Patient whose access to the puncture sites is not feasible (underlying lesions)
* Patient with allergies to local anesthetics (LA)
* Patient whose family did not give informed consent
* Patient younger than 15 years and 3 months
* Tetraplegic Patient
* Dying patients
* Patients with more than 3 different fracture sites

Ages: 183 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2014-07-31 (Actual); Study Completion 2014-07-31 (Actual)

PRIMARY OUTCOMES:
sufentanil consumption in ICU patients for sedation | up to 48 hours
  assess the interest of regional anesthesia in trauma patients with fractures members. sufentanil consumption in ICU patients for sedation (µg/kg/j)

SECONDARY OUTCOMES:
daily consumption of sufentanil | at 24 Hours
  daily consumption of sufentanil (mcg/kg/j)
daily consumption of sufentanil | 48 Hours
  daily consumption of sufentanil (mcg/kg/j)
daily consumption of sufentanil | at 72 Hours
  daily consumption of sufentanil (mcg/kg/j)
daily consumption of sufentanil | at 96 Hours
  daily consumption of sufentanil (mcg/kg/j)
daily consumption of sufentanil | at 120 Hours
  daily consumption of sufentanil (mcg/kg/j)
daily consumption of midazolam | at 24 Hours
  daily consumption of midazolam (mg/kg/j)
daily consumption of midazolam | at 48 Hours
  daily consumption of midazolam (mg/kg/j)
daily consumption of midazolam | at 72 Hours
  daily consumption of midazolam (mg/kg/j)
daily consumption of midazolam | at 96 Hours
  daily consumption of midazolam (mg/kg/j)
daily consumption of midazolam | at 120 Hours
  daily consumption of midazolam (mg/kg/j)
daily consumption of noradreline | at 24 Hours
  daily consumption of noradreline (mg/kg/j)
daily consumption of noradreline | at 48 Hours
  daily consumption of noradreline (mg/kg/j)
daily consumption of noradreline | at 72 Hours
  daily consumption of noradreline (mg/kg/j)
daily consumption of noradreline | at 96 Hours
  daily consumption of noradreline (mg/kg/j)
daily consumption of noradreline | at 120 Hours
  daily consumption of noradreline (mg/kg/j)
sedation duration | discharge, up to end of hospitalization (Follow-up up to 5 days)
  number of days between inclusion and the end of hospitalization
ventilator free days | discharge, up to end of hospitalization (Follow-up up to 5 days)
  number of days between inclusion and the end of hospitalization
duration of mechanical ventilation | discharge, up to end of hospitalization (Follow-up up to 5 days)
  number of days between inclusion and the end of hospitalization
Mechanical ventilation complication | From the third to the tenth day after inclusion
  the rate of occurrence of pneumopathy acquired under mechanical ventilation (between 3rd and 10th day of developmen

CONTACTS AND LOCATIONS:
Overall Officials: Oriane MARTINEZ, MD, Principal Investigator — Department of Anesthesia Resuscitation at the Hospital Lapeyronie
Locations (1):
- University hospital, Montpellier, France